CLINICAL TRIAL: NCT06449521
Title: A Type II Hybrid Implementation-effectiveness Study of BECOME (BEhavioral Community-based COmbined Intervention for MEntal Health and Noncommunicable Diseases) Delivered by Community Health Workers in Nepal
Brief Title: BECOME COmbined Intervention for MH & NCD Delivered by Community Health Workers in Nepal
Acronym: BECOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Possible (Other)
Collaborators: University of California, San Francisco (Other); National Institute of Mental Health (NIMH) (NIH); Ministry of Health and Population, Nepal (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: BECOMEPossible; 1R01MH133231-01 (NIH)
Record Dates: First submitted 2024-04-25; First posted 2024-06-10 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Mental Health Disorder; Non Communicable Diseases
Keywords: Mental Health; Non communicable Diseases
MeSH Terms: conditions — Mental Disorders; Noncommunicable Diseases; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study will use a stepped-wedge randomized controlled trial design. Randomization process involves sequential rolling out of the intervention in four cluster every three months. Each cluster is a ward (population ~6000), which includes one CHW and at least one basic health care clinic, with regional referrals available to higher levels of care. The 20 wards will be randomly assigned (using a random number generator) to one of five steps. All clusters begin in the control condition; every three months, four clusters will transition to the intervention condition.
  Note: The investigators have not seen better option than this one in the drop down menu above.
Masking Description: This is a stepped wedge cluster randomized controlled trial. Since participants will receive routine care when they are not receiving the BECOME intervention (which the investigators will randomly allocate using a stepped wedge fashion), the investigators will blind outcome assessors for the follow-up assessment every three months until 12 months of follow up post intervention.
  But, it's important to note that our response to masking outcome assessors cannot be recorded in above option.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm- stepped wedge implementation (Other): All participants enrolled in the study will receive intervention in a stepped wedge fashion. This means that every three months, four clusters will transition to the intervention phase until all clusters (a total of 20) in the study have received intervention. Participants will receive routine usual care when their clusters are in the control phase. This includes the Government of Nepal's (GoN) current protocols at the home/community level. CHWs will monitor for CMD and NCD symptoms and red flags every three months, provide health education, and refer individuals to health facilities.
  Interventions: Behavioral: BECOME intervention

INTERVENTIONS:
Behavioral: BECOME intervention — The intervention, BECOME, includes: a) Evidence-based stress reduction (EBSR): as recommended in the WHO mhGAP guidelines, diaphragmatic breathing and body scan will be used to manage stress and anxiety. b) Behavioral activation (BA): as recommended in the mhGAP guidelines, this evidence-based strategy will increase the time that patients spend engaging in pleasurable activities to both treat depression and increase physical activity, depending on their cognitive and physical capabilities (e.g., going to a neighbor's house for tea or walking to the local market). c) Motivational interviewing (MI): an evidence-based patient-interaction strategy that increases the patient's internal motivation to engage in healthy behaviors (e.g., quit tobacco) both to prompt change (if they are not engaging in healthy behaviors) and maintain them (if they are already engaged in healthy behaviors), as recommended by Package of Essential Noncommunicable disease interventions) PEN protocols.

SUMMARY:
Common mental health disorders (CMDs) and noncommunicable diseases (NCDs) pose significant public health challenges, especially in resource-limited settings like Nepal. The coexistence of CMDs and NCDs is prevalent, tied together by shared behavioral risk factors including stress, isolation, tobacco use, low physical activity, poor diet, and treatment non-adherence. Addressing these risk factors through behavioral interventions has the potential to positively impact both CMDs and NCDs. While the World Health Organization (WHO) recommends three behavioral interventions-evidence-based stress reduction (EBSR) for stress and anxiety, behavioral activation (BA) for depression, and motivational interviewing (MI) for healthy behaviors-availability remains scarce in low-resource settings.

This research proposes a hybrid implementation-effectiveness study of the BEhavioral Community-based COmbined Intervention for MEntal Health and Noncommunicable Diseases (BECOME) in Nepal. BECOME, delivered by community health workers (CHWs), integrates EBSR, BA, and MI to improve mental health and address NCDs. The study employs a stepped-wedge cluster randomized trial, with 20 clusters randomly assigned to five steps, starting in the control condition. Transitioning every three months, clusters gradually adopt the intervention, minimizing logistical challenges during implementation.

The study targets 600 patient participants (age 40 years and above with at least one CMD and NCD) from Bardibas and Chandragiri municipalities, involving 20 CHWs, five primary care providers (PCPs), and six health system leaders. CHWs identify potential participants, with research staff assessing eligibility, obtaining informed consent, and conducting baseline assessments using a digital REDCap tool. CHWs undergo BECOME intervention training, delivering it to consenting patient participants (30 per CHW). Quantitative data collected quarterly over 12 months will measure primary outcomes for CMDs and NCDs. Additionally, qualitative components, following the Reach Effectiveness-Adoption Implementation and Maintenance (RE-AIM) framework, include focus group discussions (FGDs) with CHWs and Key Informant Interviews (KIIs) with patient participants, PCPs, and health system leaders to assess implementation mechanisms, outcomes, and clinical impact.

The study, if successful, aims to furnish evidence and a model for implementing behavioral interventions addressing CMDs and NCDs.

DETAILED DESCRIPTION:
General Objective :

To evaluate the effectiveness and implementation of a program called BECOME on depression and/or anxiety, and two NCDs using a stepped-wedge cluster randomized trial (SWCRT) and the RE-AIM framework.

Specific Objective :

1. Assess the effectiveness of BECOME on depression and anxiety, and two NCDs (diabetes and hypertension) via a stepped-wedge cluster randomized trial.
2. Assess implementation outcomes of BECOME using the RE-AIM framework at the patient, provider, and health system levels
3. Conduct a comprehensive costing analysis to provide strategic inputs to support long-term scale up of BECOME.

Study Variables Dependent variable; Primary outcome: depression and anxiety severity, Secondary outcome: Diabetes (as measured by fasting plasma glucose) and hypertension (as measured by systolic and diastolic blood pressure) Independent variable; Demographics (for example, age, sex) Stress, Isolation and withdrawal, Quality of Life, Tobacco Use, Diet Quality, Physical activity, Medication and follow up adherence, Environmental factors- access to care (community-based and higher intensity clinical care), social support, life style.

Research Method : mixed

Study sites : Bardibas and Chandragiri municipalities, Nepal

Specify type of Study This study is a type-II hybrid effectiveness- implementation study. The study will use a stepped-wedge randomized controlled trial design.

Study Population

Patient Participants: Individuals who are 40 years or above residing in Chandragiri and Bardibas Municipalities who have at least one NCD (hypertension and/or diabetes) and one Mental Health (depression and/or anxiety), and who give consent for the study participation.

Community health workers: Community health workers who are working in Chandragiri and Bardibas municipalities under the government pilot program following community health program guidelines 2078 endorsed by the Ministry of Health and Population. They are the community health nurses employed by municipalities. They are the trusted local member of the community who are trained and regularly supported and monitored by their supervisors. They work full-time and get a monthly salary for their service/work.

Primary care providers and health system leaders: who are working either in the health facilities of Chandragiri and Bardibas municipalities, municipal health office, and relevant stakeholders who are contributing to the community health program in different capacities.

Sampling unit

Since this is a stepped wedge cluster randomized controlled trial, investigators will use the cluster as our sampling unit while implementing the study.

Sample size

631 Participants; 20 CHWs; 5 Primary care providers; 6 Health system leaders

Description of study design:

The is a type-II hybrid effectiveness-implementation study design. The goal of the effectiveness aim is to evaluate the impact of the BECOME intervention against usual care while the implementation aim focuses on understanding the process of implementing the intervention in a real-world setting. Additionally, the study will conduct a comprehensive costing analysis to provide strategic inputs to support the long-term scale-up of BECOME.

The study will use a stepped-wedge cluster randomized controlled trial design. In this design, 20 clusters (wards) will be randomly assigned to one of five steps, with all clusters starting in the control phase prior to receiving the intervention. Every three months, four clusters will transition to the intervention condition, while the remaining clusters will remain in the control condition. This design allows for a gradual rollout of the intervention, which can help minimize the impact of any learning curves or logistical challenges that may arise during implementation.

The study will use an open cohort design, which means that enrollment will be kept open while the intervention is being offered. This approach helps to reflect real-world conditions and can compensate for attrition and for participants who may no longer meet the eligibility criteria when their cluster transitions to the treatment phase. By using this design, the study can capture the dynamic nature of the intervention and better understand its impact over time.

Overall, this study aims to evaluate the effectiveness and implementation of the BECOME intervention, as well as provide insights into the costs associated with implementing the intervention in a real-world setting. By using a stepped-wedge cluster randomized controlled trial design and an open cohort design, the study can capture a comprehensive picture of the intervention's impact and implementation process.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women age ≥ 40 years
* Living in the target wards with no intention of leaving in the next 2.5 yrs
* Anxiety (HSCL-25 anxiety subscale score ≥1.75) and/or Depression (HSCL-25 depression subscale score ≥1.75)
* At least one Non-communicable disease (NCD) based on WHO PEN criteria; either Hypertension (HTN) (SBP ≥130mmHg and/or DBP ≥80mmHg) and/or Diabetes Mellitus (DM) (fasting plasma glucose (FPG) ≥126mg/dl or random plasma glucose ≥200mg/dl)

Exclusion Criteria:

* Significant cognitive problems/disability
* Pregnant women
* Postpartum (≤6 weeks) women

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Lower Mean Hopkins Symptom Checklist-25 (HSCL-25) score | First in baseline assessment and then every 3 months up to 12 months from the start of BECOME intervention.
  The Hopkins Symptom Checklist-25 is a measure of symptoms of anxiety and depression. This instrument consists of two different subscales; one for anxiety symptoms and the other for depression. The scale for each question includes four response categories ("Not at all," "A little," "Quite a bit," and "Extremely," rated 1 to 4, respectively). The scores range from 1 to 4. Higher score shows higher severity of anxiety and depression symptoms.

SECONDARY OUTCOMES:
Mean systolic blood pressure in millimeters of mercury (mmHg) | First in baseline assessment and then every 3 months up to 12 months from the start of BECOME intervention.
  The two consecutive measurements of systolic blood pressure (SBP) measured at the interval of 3 minutes will be used to calculate the mean systolic blood pressure. Portable digital blood pressure machine will be used for the measurement.
Mean diastolic blood pressure in millimeters of mercury (mmHg) | First in baseline assessment and then every 3 months up to 12 months from the start of BECOME intervention.
  The two consecutive measurements of diastolic blood pressure (DBP) measured at the interval of 3 minutes will be used to calculate the mean diastolic blood pressure. Portable digital blood pressure machine will be used for the measurement.
Fasting plasma glucose in milligrams per deciliter (mg/dL) | First in baseline assessment and then every 3 months up to 12 months from the start of BECOME intervention.
  Fasting plasma glucose will be measured by portable glucometer machine.

CONTACTS AND LOCATIONS:
Overall Officials: Bibhav Acharya, MD, Principal Investigator — University of California, San Francisco; Sabitri Sapkota Devkota, PhD, Principal Investigator — Possible
Locations (1):
- Possible, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share ONLY the de identified data through NIH designated data repositories consistent with data sharing under the NIH GDS policy. The investigators will include the clinical data of those research participants who will provide consent for sharing their data.
Supporting Information: CSR
Time Frame: Final submission and release of the study data will occur approximately 12 months following the end of the trial, and within the award period. Study data deposited in the repository will be available to the research community in perpetuity. Datasets underlying methodological publications will be shared at or prior to initial publication date.
Access Criteria: The investigators will share ONLY the deidentified data through NIH designated data repositories consistent with data sharing under the NIH GDS policy. The investigators will include the clinical data of those research participants who will provide consent for sharing their data.

REFERENCES:
- [Background] mhGAP Intervention Guide for Mental, Neurological and Substance Use Disorders in Non-Specialized Health Settings: Mental Health Gap Action Programme (mhGAP): Version 2.0. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK390828/ PMID 27786430
- [Background] Hettema JE, Hendricks PS. Motivational interviewing for smoking cessation: a meta-analytic review. J Consult Clin Psychol. 2010 Dec;78(6):868-84. doi: 10.1037/a0021498. PMID 21114344
- [Background] Lai DT, Cahill K, Qin Y, Tang JL. Motivational interviewing for smoking cessation. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD006936. doi: 10.1002/14651858.CD006936.pub2. PMID 20091612
- [Background] Li Z, Chen Q, Yan J, Liang W, Wong WCW. Effectiveness of motivational interviewing on improving Care for Patients with type 2 diabetes in China: A randomized controlled trial. BMC Health Serv Res. 2020 Jan 23;20(1):57. doi: 10.1186/s12913-019-4776-8. PMID 31973759
- [Background] Heckman CJ, Egleston BL, Hofmann MT. Efficacy of motivational interviewing for smoking cessation: a systematic review and meta-analysis. Tob Control. 2010 Oct;19(5):410-6. doi: 10.1136/tc.2009.033175. Epub 2010 Jul 30. PMID 20675688
- [Background] Lundahl B, Moleni T, Burke BL, Butters R, Tollefson D, Butler C, Rollnick S. Motivational interviewing in medical care settings: a systematic review and meta-analysis of randomized controlled trials. Patient Educ Couns. 2013 Nov;93(2):157-68. doi: 10.1016/j.pec.2013.07.012. Epub 2013 Aug 1. PMID 24001658
- [Background] Sayegh CS, Huey SJ, Zara EJ, Jhaveri K. Follow-up treatment effects of contingency management and motivational interviewing on substance use: A meta-analysis. Psychol Addict Behav. 2017 Jun;31(4):403-414. doi: 10.1037/adb0000277. Epub 2017 Apr 24. PMID 28437121
- [Background] Anthonisen NR, Skeans MA, Wise RA, Manfreda J, Kanner RE, Connett JE; Lung Health Study Research Group. The effects of a smoking cessation intervention on 14.5-year mortality: a randomized clinical trial. Ann Intern Med. 2005 Feb 15;142(4):233-9. doi: 10.7326/0003-4819-142-4-200502150-00005. PMID 15710956
- [Derived] Sigdel K, Nepal J, Shrestha A, Rai B, Yogi B, Schillinger D, Sharma D, Prajapati D, Heylen E, Niraula HK, Shrestha J, Dhimal M, Sah NK, Baral PP, Limbu P, Nepal P, Paudel P, Nepali S, Poudel S, Joshi S, Tiwari S, Shrestha S, Sapkota S, Acharya B. A type II hybrid implementation-effectiveness study of the BECOME intervention: integrating Behavioral Community-Based Approaches for Mental Health and Non-Communicable Diseases delivered by community health workers-study protocol for a stepped wedge cluster randomized controlled trial. Trials. 2026 Jan 24. doi: 10.1186/s13063-026-09457-1. Online ahead of print. PMID 41580851